CLINICAL TRIAL: NCT06372314
Title: Isoleucine, Leucine, Valine and Tryptophan Requirements in Total Parenteral Nutrition (TPN) Fed Neonates
Brief Title: Isoleucine, Leucine, Valine and Tryptophan Requirements in TPN Fed Neonates
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Glenda Courtney-Martin, Principal Investigator, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1000081221
Record Dates: First submitted 2024-04-15; First posted 2024-04-18 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Stable Neonates Receiving Total Parenteral Nutrition (TPN)
Keywords: Neonates, Total pareteral nutrition (TPN), Isoleucine, Leucine, Valine, Tryptophan
MeSH Terms: interventions — Parenteral Nutrition, Total

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Isoleucine, leucine, valine, tryptophan requirement (Experimental): isoleucine, leucine, valine and tryptophan intakes will be varied in the TPN solutions to study the requirements for each of these amino acids in neonates that are TPN fed.
  Interventions: Drug: Total parenteral nutrition (TPN): this is total nutrition provided by central vein.

INTERVENTIONS:
Drug: Total parenteral nutrition (TPN): this is total nutrition provided by central vein. — isoleucine, leucine, valine and tryptophan intakes will be varied in the TPN solutions to study the requirements for each of these amino acids in neonates that are TPN fed.

SUMMARY:
This project will be conducted in 2 hospitals in Brazil to assess the requirements for four essential amino acids in TPN fed neonates. Using the Carbon Oxidation method (indicator amino oxidation and direct amino acid oxidation method), the investigators will determine the requirement of each of the 4 amino acids.

The investigators will determine the requirement for Isoleucine, Leucine, Valine and Tryptophan. The investigators will recruit 18- 20 babies per amino acid study. Breath and urine samples will be collected to determine the oxidation of the indicator amino acid. The response of the indicator amino acid to changes in intake of the test amino acid (isoleucine, leucine, valine and tryptophan) will be analyzed by bi-phase linear mixed effect model to determine the breakpoint or mean requirement for each amino acid. It is hypothesized that the requirement for isoleucine, leucine, valine and tryptophan will be at least 50% lower than what is currently available in commercial solutions used for TPN feeding of neonates.

DETAILED DESCRIPTION:
The study is based on the carbon oxidation protocol. Each baby will receive one or two levels of either isoleucine or leucine or valine or tryptophan. Each level will be assessed over a two- day period.

On day 1: each baby will receive a standard pediatric amino acid solution, Primene used in the NICU and L-[1-13C]Na Bicarbonate will be given to measure carbon dioxide production.

On day 2: he/she will receive the appropriate TPN Test Solution made up of the appropriate Bulk Amino Acid solution (for Isoleucine/ Leucine/ Valine/ Tryptophan Studies) with a different amount of the amino acid being investigated. To see how these amino acids are used in the body the investigators will add a small amount (calculated based on the body weight of the baby) of the amino acid L-[1-13C]phenylalanine to the amino acid solution. Breath and urine will be collected from the baby to study the oxidation of the L -[1-13C]phenylalanine. The investigators will take 2 x 0.75 ml blood to measure plasma amino acid concentration. The investigators will aim to coordinate blood taking with routine blood work done for clinical monitoring.

ELIGIBILITY:
Inclusion Criteria:

1. Stable preterm babies that are growing and fully TPN fed (at least 90% of calories and protein).
2. TPN providing adequate calories and protein as determined by attending physician and dietitian.
3. Babies born ≥ 28 weeks gestation,
4. ≤ 28 days chronological age at the time of the study,
5. Birth weight and length appropriate for gestational age,
6. Medically stable as determined by normal blood results and lack of a fever or infection,
7. At least 3 days after surgery, if the baby had a surgery

Exclusion Criteria:

1. Babies on mechanical ventilation, on low flow oxygen and CPAP.
2. Small for gestational age,
3. On medications known to affect protein and amino acid metabolism,
4. Documented infection, fever
5. Unstable medical condition
6. Receiving enteral feeding providing > 10% of protein intake

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Amino acid oxidation using a labelled amino acid. | 48 hrs
  Breath samples will be collected and analyzed to determine the amount ofamino acid oxidized. This will be used to determine the amount retained inthe body and therefore the amount that is required for protein synthesis.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de Caridade Dr. Astrogildo de Azevedo, and University Hospital of Santa Maria, Santa Maria, Brazil, Santa Maria, Brazil

IPD SHARING:
Plan to Share IPD: No